CLINICAL TRIAL: NCT07069374
Title: Wellness, Intervention Strategies and HIV Care
Acronym: WISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K01DA056306 (NIH); K01DA056306 (NIH)
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HIV; Substance Use Disorder (SUD)
Keywords: HIV; Substance Use; Risk Reduction; Behavioral Intervention; Public Health; Intervention Program
MeSH Terms: conditions — Substance-Related Disorders; Risk Reduction Behavior | interventions — Health; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants in this arm will attend a structured, group-based behavioral support program consisting of five weekly sessions. The intervention is designed for individuals living with HIV who use substances. It focuses on strategies for managing stress, reducing barriers to care, and improving engagement in HIV-related health services and overall wellness.
  Interventions: Behavioral: Wellness, Intervention Strategies and HIV Care (WISH)
- Control Arm (Placebo Comparator): Participants in this arm will attend five weekly group-based sessions where non-intervention-related movies are shown. This condition is intended to control for time and group exposure without delivering active behavioral content related to the study outcomes.
  Interventions: Behavioral: Movie Night Club - Attention and Time Matched Control

INTERVENTIONS:
Behavioral: Wellness, Intervention Strategies and HIV Care (WISH) — A structured behavioral group program consisting of five weekly sessions, each approximately 60-90 minutes in length. The intervention is designed for individuals living with HIV who use substances and focuses on: managing stress, addressing barriers to care, and enhancing engagement with HIV-related health services. Sessions are delivered in a small-group format and facilitated by trained staff using a manualized curriculum.
  Arms: Intervention Arm
Behavioral: Movie Night Club - Attention and Time Matched Control — Weekly 90-minute group sessions over 5 weeks in which participants watch non-therapeutic, neutral-content movies in a group setting. Sessions are facilitated to control for social interaction and time spent in a structured group environment but do not include any therapeutic content.
  Arms: Control Arm

SUMMARY:
This is a pilot trial designed to assess the feasibility and acceptability of an intervention aimed at improving adherence to antiretroviral therapy (ART), viral suppression, and engagement in HIV care. The intervention will address behavioral coping strategies, HIV care engagement behaviors, and substance use management.

ELIGIBILITY:
Inclusion Criteria:

• Participants must:

* Be at least 18 years of age
* Self-report biological characteristics consistent with the population under study
* Be HIV-positive
* Report use of at least one of the following substances in the last 90 days:

  * Cannabis
  * Methamphetamine
  * Cocaine/crack
  * Cocaine
  * Heroin
  * Non-prescribed opioids (e.g., fentanyl, morphine)
  * Ecstasy
  * Phencyclidine (PCP)
  * Psychedelics (e.g., Lysergic acid diethylamide, mescaline, ketamine)
  * Poppers (alkyl nitrites)
  * Non-prescribed benzodiazepines (e.g., Valium, Xanax, Klonopin, Librium)
  * Barbiturates
* Be English-speaking
* Be able and willing to provide informed consent

Exclusion Criteria:

* Evidence of severe cognitive impairment or active psychosis that may impede ability to provide fully informed consent, determined by the research assistants and clinical supervisor(s)
* The research staff are trained on guidelines for identifying participants who exhibit signs of inability to meaningfully participate or provide consent due to mental illness or impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The Client Satisfaction Questionnaire (CSQ-8) | 6 Months
  The Client Satisfaction Questionnaire-8 (CSQ-8) consists of eight items, each rated on a 4-point Likert scale. Total scores range from 8 to 32, with higher scores indicating greater satisfaction with the services received.
Acceptability of Intervention Measure (AIM) | 5 Weeks
  The AIM consists of 4 items rated on a 5-point Likert scale, ranging from 1 (completely disagree) to 5 (completely agree). Total scores range from 4 to 20, with higher scores indicating greater acceptability of the intervention.
Participant Retention Rate | 5 Weeks
  The percentage of participants who complete the intervention protocol. Calculated as (number of participants completing the study ÷ number enrolled) × 100%. A retention rate of ≥70% will indicate protocol adherence feasibility.
Participant Enrollment Rate | 6 Months
  The proportion of participants enrolled out of those screened for eligibility. This will be calculated as (number enrolled ÷ number screened) × 100%. An enrollment rate of ≥70% will be considered feasible, based on clinical standards in the literature.
Number of Staff Members Required for Study Implementation | 6 Months
  Total number of staff members involved in intervention delivery and data collection, documented throughout the pilot period.
Feasibility of Intervention Measure (FIM) | 5 Weeks
  The FIM includes 4 items rated on a 5-point Likert scale, from 1 (completely disagree) to 5 (completely agree). Total scores range from 4 to 20, with higher scores indicating greater perceived feasibility of the intervention.

SECONDARY OUTCOMES:
Binary Measure of Optimal Adherence to ART (≥85%) | 6 Months
  Adherence will be assessed using participant self-report over the prior three months. A binary outcome will be calculated: participants with an adherence rate of 85% or higher will be classified as "optimal adherence," and those below 85% as "non-optimal adherence." This measure reflects adherence to the assigned intervention.
Binary Measure of HIV Viral Suppression (<200 copies/mL) | Baseline, 3 months, and 6 months
  HIV viral load will be measured using plasma HIV RNA nucleic acid tests. Viral suppression is defined as <200 copies/mL, and non-suppression as >200 copies/mL, in accordance with Department of Health and Human Services and AIDS Clinical Trials Group guidelines.
Cumulative Adherence to TDF/TAF as Measured by Drug Concentration in Hair Samples | 6 Months
  Cumulative adherence will be assessed by quantifying levels of tenofovir disoproxil fumarate (TDF) and tenofovir alafenamide (TAF) in hair samples. Drug concentrations will be measured using validated LC-MS/MS assays. Higher drug levels indicate greater cumulative adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer P Jain, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Oakland MWCCS Site Office, Oakland, California
  - SF MWCCS Site Office, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available beginning 12 months after the completion of data collection through a secure, NIH-approved data repository. Access will be granted to qualified researchers who provide a data use request and comply with data sharing agreements. Shared data will not include direct identifiers and will be limited to information consistent with participant consent.
Time Frame: IPD will be available beginning 12 months after the primary completion date of the study. IPD will be available for up to 5 years after the initial release date, or longer if the repository's policies permit extended access.
Access Criteria: De-identified individual participant data (IPD) and supporting documentation (such as the data dictionary) will be made available to qualified researchers whose proposed use of the data has been approved by the study PI. Approved users will be granted access through a secure NIH-designated repository, contingent upon completion of a data use agreement. Shared data will include baseline characteristics, outcome measures, and other variables as outlined in the data management and sharing plan, excluding any direct identifiers.